CLINICAL TRIAL: NCT04490616
Title: EFFECTS of RTMS TREATMENT on SOCIAL COGNITION DYSFUNCTIONS in MILD COGNITIVE IMPAIRMENT: an PROSPECTIVE, DOUBLE-BINDING, RANDOMIZED, SINGLE CENTRE, EXPLORATIVE STUDY
Brief Title: TMS Treatment of Social Cognition Skills in Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedale Regionale di Lugano (Other)
Responsible Party: Principal Investigator, Leonardo Sacco, Principal Investigator, Ospedale Regionale di Lugano
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-00434/CE 3594
Record Dates: First submitted 2020-07-10; First posted 2020-07-29 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2023-10

CONDITIONS: Mild Cognitive Impairment
Keywords: ripetitive transcranial magnetic stimulation treatment; social cognition; theory of mind; empathy; social perception; social behavior
MeSH Terms: conditions — Cognitive Dysfunction; Social Behavior

STUDY DESIGN:
Intervention Model Description: In the project will be applied a two-site repetitive transcranial magnetic stimulation (rTMS) stimulation.
  MCI patients that obtained a score ≤ 10 percentiles, at least one performance/domain of social cognition assessment will be considered impaired at social cognition abilities. In the same day of cognitive-behavioral assessment, patients will be randomly assigned to one of the two groups:
  1) RR-Gr received 4 weeks of rTMS stimulation of the RTPJ and MPFC; (2) SR-Gr received of the RTPJ and MPFC sham stimulation during the first 2 weeks followed by 2 weeks of real stimulation. Each week of rTMS treatment consisted of five sessions. This paradigm has proven to be effective for improve cognitive performances in AD patients. In the sham condition, a sham coil will be used.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RR-GR (Experimental): MCI patients with social cognition deficits will receive 4 weeks of rTMS stimulation
  Interventions: Other: rTMS treatment
- SR-GR (Other): MCI patients with social cognition deficits will receive 2 weeks of placebo treatment, followed by 2 weeks of real rTMS stimulation
  Interventions: Other: rTMS treatment

INTERVENTIONS:
Other: rTMS treatment — A two-site rTMS stimulation delivered by a Magstim unit featuring a double 70 mm cooled coil will be applied.
  MCI patients will be randomly assigned to one of the two study groups:
  1. RR-Gr will receive 4 weeks of rTMS stimulation of the right temporo-parietal junction (RTPJ) and medial prefrontal cortex (MPFC);
  2. PL-Gr will receive sham stimulation of the RTPJ and MPFC during the first 2 weeks followed by 2 weeks of real stimulation. Each week of rTMS treatment will consist of five sessions (50 min, one per day).
  For each area target, a total of 2000 pulses at 20Hz, 3-s train duration, and 28-s inter-train interval at 100% motor threshold (MT) will be delivered per session. A fixed intensity of MT will ensure a more consistent spatial spread of TMS effects in subjects' brains not influenced by differences in individual MT. In the sham condition, a sham coil will be used.
  Each session lasted for about 60 min including time for set up and 50 min of stimulation.

SUMMARY:
Social cognitive abilities are impaired in around 17% of subjects with mild cognitive impairment (MCI), and might not reflect upon functional status. Compared to healthy controls, MCI showed impairments in theory of mind (ToM) and facial emotion recognition. Moreover, in amnesic MCI patients, reduced ToM ability appears to be correlated with worse performances at several cognitive performances. These findings, in agreement with previous evidence, confirm that impaired social cognition might occur prior to dementia: typically elderly start to show impairment in the complex ToM levels, which is found also in MCI patients and proceeds further in AD patients. Thus, the treatment of these aspects has the potential to influence the trajectory of neurodegeneration. In the last decade, it has been increasingly evident the effectiveness of active stimulation of brain regions with repetitive transcranial magnetic stimulation (rTMS), to improve cognitive and functional performances in patients with dementia.

On the other hand, brain imaging techniques and TMS stimulations have identified two main areas responsible for human social cognition- the medial prefrontal cortex (MPFC) and the right temporo-parietal junction (RTPJ).

In this project, we hypothesized that an improvement of social cognition skills may be obtained in MCI patients by using the rTMS on two main areas responsible for human social cognition- the medial prefrontal cortex (MPFC) and the right temporoparietal junction (RTPJ). Moreover, it expects that rTMS treatment may also contribute to improving cognitive abilities and neuropsychiatric aspects partially modulated by the same networks stimulated.

DETAILED DESCRIPTION:
This is a prospective, double-binding, cross-sectional, randomized, sham-controlled, and single-center project aimed to investigate the effect of rTMS treatment of social cognition abilities in MCI subjects at 2 and 4 weeks, and after 8 weeks from baseline.

All patients will be recruited at Clinical Neuroscience Institute, Department of Neurology, Regional Civic Hospital, Lugan; Department of Geriatric Italian Hospital Viganello; and Department of Geriatric, Beata Vergine Hospital Mendrisio; Southern Switzerland, Switzerland.

Primary objective:

1. To investigate whether the application of high-frequency rTMS, for 2 or 4 weeks, to the RPTJ and MPFC resulted in social cognitive improvements.

Secondary objectives:

1. To verify whether the social cognition benefits previously recorded might persist after 8 weeks the end of the stimulation, with a major benefit with a longer rTMS application (4 weeks).
2. To investigate whether the application of high-frequency rTMS, at 2 weeks or 4 weeks, to the RPTJ and MPFC contributes to improve cognitive functions as well as neuropsychiatric (depression) and functional aspects.
3. To verify whether the cognitive functions, neuropsychiatric aspect, and functional benefits previously recorded persist after the end of the rTMS stimulation.

Primary analysis: To investigate the behavioral effects induced by the rTMS protocol after 2 and 4 weeks of daily stimulation on social cognition skills, executive/attentive functions, neuropsychiatric and functional aspects will be used a mixed-model ANOVA, considering the group as a between-subjects factor, and time as a within-subject factor.

Secondary Analyses: To investigate the direct or mediated rTMS effect on social cognition skills, a multivariate linear regression analysis will be done for each social cognition measure (ToM, empathy, social perception, social behavior) changes after rTMS treatment at 2 and 4 weeks as the dependent factor, separately, and appropriate screening/baseline dependent variables and rTMS groups as independent factors.

The evaluation and treatment of social cognition alterations in subjects with MCI can be useful for two main aspects: first, the mild cognitive and behavior impairment of these subjects favor a better answer at the treatment, both at the behavioral level and in terms of brain structural and functional response; second, treatment of these abilities in MCI population might retard the conversion to dementia. More importantly, the detection of predominant social cognition alteration in early phases of cognitive decline might be potentially helpful to differentiate individuals who will develop frontotemporal dementia. Therefore, it is important to investigate and define a treatment protocol to limit social cognition disturbances in MCI.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 50 to 85 years old, inclusive, at the time of informed consent;
* Must have at least 5 years of education or work experience to exclude mental deficits other than MCI;
* Must meet Petersen's criteria for mild cognitive impairment, and must have:
* Clinical dementia rating global score of 0.5;
* Mini-Mental State Examination score between 24 and 30;
* Must have a score ≥ 26.5 at Token test to ensure that subjects have the ability to understand the instructions and procedures;
* Must have a score < 29 at Beck Depression Inventory to exclude major depression that could compromise the patient's ability to engage in the study;
* Apart from a clinical diagnosis of MCI, the subject must be in good health;
* Must be on stable dose of antidepressant (if applicable) for at least 2 months prior to the enrolment.

Exclusion Criteria:

* Any uncontrolled medical or neurological/neurodegenerative condition (other than MCI);
* Clinical significant unstable psychiatric illness requiring treatment with neuroleptic;
* Transient ischemic attack, stroke, or any unexplained loss of consciousness or severe ongoing stressor within 1 year prior to screening;
* History of seizure within10 years prior to screening;
* Recent history of alcohol or substance abuse or use of cannabinoids;
* Any other medical conditions that are not stable or controlled, or could affect the subject's safety or interfere with the study assessments and treatment;
* Contraindication to having TMS treatment;
* Inability to understand the purpose of the study or to comply with study requirements.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-02-11 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Comparison of Deceptive Box Task score | Week 2
  (5 items). Minimum value=0, maximum value=5. A higher score means a better outcome.
Comparison of Look-prediction/say-prediction test score | Week 2
  (5 items). Minimum value=0, maximum value=5. A higher score means a better outcome.
Comparison of Empathy Quotient score | Week 2
  (60 items). Minimum value=0, maximum value=80. A higher score means a better outcome.
Comparison of Ekman 60 test score | Week 2
  (60 b/w pictures). Minimum value=0, maximum value=60. Higher score means a better outcome.
Comparison of Frontal Behavioral Inventory score | Week 2
  (24 items). Minimum value=0, maximum value=69. Higher score means a worse outcome.
Comparison of Deceptive Box Task score | Week 4
  (5 items). Minimum value=0, maximum value=5. A higher score means a better outcome.
Comparison of Look-prediction/say-prediction test | Week 4
  (5 items). Minimum value=0, maximum value=5. A higher score means a better outcome.
Comparison of Empathy Quotient score | Week 4
  (60 items). Minimum value=0, maximum value=80. A higher score means a better outcome.
Comparison of Ekman 60 test score | Week 4
  (60 b/w pictures). Minimum value=0, maximum value=60. Higher score means a better outcome.
Comparison of Frontal Behavioral Inventory score | Week 4
  (24 items). Minimum value=0, maximum value=69. Higher score means a worse outcome.

SECONDARY OUTCOMES:
Changes from baseline in Deceptive Box Task Test. | Week 12
  (5 items). Minimum value=0, maximum value=5. A higher score means a better outcome.
Changes from baseline in Look/say Test | Week 12
  (5 items). Minimum value=0, maximum value=5. A higher score means a better outcome.
Changes from baseline in Empathy Quotient scale | Week 12
  (60 items). Minimum value=0, maximum value=80. A higher score means a better outcome.
Changes from baseline in Ekman 60 Test | Week 12
  (60 b/w pictures). Minimum value=0, maximum value=60. Higher score means a better outcome.
Changes from baseline in Frontal Behavioral Inventory | Week 12
  (24 items). Minimum value=0, maximum value=69. Higher score means a worse outcome.
Comparison Montreal Cognitive Assessment | through study completion, an average of 12 weeks
  (30 items). Minimum value=0, maximum value=30. Higher score means a better outcome.
Comparison of Geriatric Depression Scale score | through study completion, an average of 12 weeks
  (30 items). Minimum value=0, maximum value=30. Higher score means a better outcome.
Comparison of Euroquol-5 dimensions score | athrough study completion, an average of 12 weeks
  (visual analogue scale with 100-point scale). Minimum value=0, maximum value=100. Higher score means a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo Sacco, Dr, Principal Investigator — +41 091 811 6921
Locations (1):
- Neurocentro della Svizzera italiana,Ospedale Regionale di Lugano, Lugano, Canton Ticino, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baumgardner DJ, Christopherson A, Momont S. Chlamydia in pregnant women: southeastern Wisconsin. Wis Med J. 1989 Sep;88(9):12-5. PMID 2588649
- [Background] Wondra JD, Ellsworth PC. An appraisal theory of empathy and other vicarious emotional experiences. Psychol Rev. 2015 Jul;122(3):411-28. doi: 10.1037/a0039252. Epub 2015 May 11. PMID 25961468
- [Background] Apperly IA, Samson D, Chiavarino C, Humphreys GW. Frontal and temporo-parietal lobe contributions to theory of mind: neuropsychological evidence from a false-belief task with reduced language and executive demands. J Cogn Neurosci. 2004 Dec;16(10):1773-84. doi: 10.1162/0898929042947928. PMID 15701227
- [Background] Wood JN, Knutson KM, Grafman J. Psychological structure and neural correlates of event knowledge. Cereb Cortex. 2005 Aug;15(8):1155-61. doi: 10.1093/cercor/bhh215. Epub 2004 Nov 24. PMID 15563720
- [Background] Van Overwalle F. Social cognition and the brain: a meta-analysis. Hum Brain Mapp. 2009 Mar;30(3):829-58. doi: 10.1002/hbm.20547. PMID 18381770
- [Background] Amodio DM, Frith CD. Meeting of minds: the medial frontal cortex and social cognition. Nat Rev Neurosci. 2006 Apr;7(4):268-77. doi: 10.1038/nrn1884. PMID 16552413
- [Background] Cabeza R, Ciaramelli E, Moscovitch M. Cognitive contributions of the ventral parietal cortex: an integrative theoretical account. Trends Cogn Sci. 2012 Jun;16(6):338-52. doi: 10.1016/j.tics.2012.04.008. Epub 2012 May 19. PMID 22609315
- [Background] Dodich A, Cerami C, Crespi C, Canessa N, Lettieri G, Iannaccone S, Marcone A, Cappa SF, Cacioppo JT. Differential Impairment of Cognitive and Affective Mentalizing Abilities in Neurodegenerative Dementias: Evidence from Behavioral Variant of Frontotemporal Dementia, Alzheimer's Disease, and Mild Cognitive Impairment. J Alzheimers Dis. 2016;50(4):1011-22. doi: 10.3233/JAD-150605. PMID 26836153
- [Background] Freedman M, Binns MA, Black SE, Murphy C, Stuss DT. Theory of mind and recognition of facial emotion in dementia: challenge to current concepts. Alzheimer Dis Assoc Disord. 2013 Jan-Mar;27(1):56-61. doi: 10.1097/WAD.0b013e31824ea5db. PMID 22407224
- [Background] Padala PR, Padala KP, Lensing SY, Jackson AN, Hunter CR, Parkes CM, Dennis RA, Bopp MM, Caceda R, Mennemeier MS, Roberson PK, Sullivan DH. Repetitive transcranial magnetic stimulation for apathy in mild cognitive impairment: A double-blind, randomized, sham-controlled, cross-over pilot study. Psychiatry Res. 2018 Mar;261:312-318. doi: 10.1016/j.psychres.2017.12.063. Epub 2018 Jan 5. PMID 29331848
- [Background] Ferrari C, Vecchi T, Todorov A, Cattaneo Z. Interfering with activity in the dorsomedial prefrontal cortex via TMS affects social impressions updating. Cogn Affect Behav Neurosci. 2016 Aug;16(4):626-34. doi: 10.3758/s13415-016-0419-2. PMID 27012713
- [Background] Cotelli M, Manenti R, Cappa SF, Zanetti O, Miniussi C. Transcranial magnetic stimulation improves naming in Alzheimer disease patients at different stages of cognitive decline. Eur J Neurol. 2008 Dec;15(12):1286-92. doi: 10.1111/j.1468-1331.2008.02202.x. PMID 19049544
- [Background] Cotelli M, Calabria M, Zanetti O. Cognitive rehabilitation in Alzheimer's Disease. Aging Clin Exp Res. 2006 Apr;18(2):141-3. doi: 10.1007/BF03327429. PMID 16702783
- [Derived] Riccitelli GC, Beeching F, Lecchi A, Ongaro G, Pertoldi W, Kaelin-Lang A, Sacco L. Enhancing Social Cognition in Mild Cognitive Impairment with Non-Invasive Brain Stimulation: A Randomized Clinical Trial. Neurorehabil Neural Repair. 2025 Dec;39(12):972-982. doi: 10.1177/15459683251360731. Epub 2025 Aug 21. PMID 40838395